CLINICAL TRIAL: NCT03611088
Title: Effect of Kangaroo Position on Electromyographic Activity, Macrocirculation and Microcirculation of Preterm Newborns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Rafael Moura Miranda, Principal Investigator, Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 69847917.7.0000.5201
Record Dates: First submitted 2018-07-16; First posted 2018-08-02 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Kangaroo Mother Care Method
Keywords: Child Development; Kangaroo Mother Care Method; Electromyography; Microcirculation; Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newborns submitted to Kangaroo Position. (Experimental)
  Interventions: Other: Kangaroo Position.
- Newborns not submitted to Kangaroo Position. (No Intervention)

INTERVENTIONS:
Other: Kangaroo Position. — The kangaroo position - the newborn is positioned in the adult's breasts, face down, should be dressed in light clothes and wrapped in a flexible cloth.
  Arms: Newborns submitted to Kangaroo Position.

SUMMARY:
Growing evidences indicates that the Kangaroo Mother Method is associated with health benefits for the child and her mother. Improvements have been found in physiological parameters of the preterm infants assisted by the method. Some of them are the reduction of the heart rate and respiratory, as well as the increase of the body temperature and of the arterial saturation of oxygen. More recently, it has been observed that children submitted to the method present an improvement in muscle tone, by the increase in the electromyographic activity of the biceps brachii and hamstrings. These physiological changes can result in benefits for the child, with a positive influence on their development.

It is well established that the preterm newborn has an important circulatory vulnerability, since the transition from fetal life to extrauterine life is a complex process in which the major changes are concentrated in the cardiovascular system and occur during the first Hours after birth accompanied by important consequences in physiological parameters, such as systemic vascular resistance, heart rate and blood flow in the organs. Therefore, global hemodynamic parameters have been studied in premature infants, especially after some intervention. It is worth noting, however, that these global parameters such as blood pressure, heart rate and arterial oxygen saturation do not reflect the existence of adequate tissue oxygenation, since they are macrocirculatory and non-microcirculatory parameters. In order to obtain reliable signals on tissue oxygenation, it is essential to study the microcirculation.

To further explore the effects that Kangaroo Position promotes on the physiological aspects of the newborn, especially on hemodynamic parameters, we consider it important to study aspects that may, in fact, represent an adequate tissue oxygenation. Therefore, the objective of this study is to evaluate the effect of Kangaroo Position in the electromyographic activity and on hemodynamic parameters, by means of microcirculation/macrocirculation measurements.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns with gestational ages older or equal than 27 and less than 37 completed weeks of gestation (Ballard Method)
* Preterm newborns hospitalized at Instituto de Medicina Integral Prof. Fernando Figueira (IMIP) with a corrected age less than 37 weeks at the moment of the evaluation
* Preterm newborns who were not submitted to the Kangaroo Position previously.

Exclusion Criteria:

* Apgar less than 7 in the 5''
* Previous history of intracranial hemorrhage (diagnosed by ultrasonography and recorded in the medical record)
* Previous convulsion history
* Congenital infection
* Infections of the central nervous system (meningitis or encephalitis)
* Malformations in the central nervous system
* Congenital cardiopaths
* Trauma during delivery
* Gastroesophageal reflux disease
* Phototherapy and anemia

Ages: 27 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
Electromyographic activity | 1 minute
  Represented by the recording of the myoelectric signal captured through the electromyographic analysis, analyzed in Root Mean Square (RMS) and measured in microvolts.
oxygen artery saturation | 1 minute
  Represented by the macrocirculation variables
heart rate | 1 minute
  Represented by the macrocirculation variables
tissue oxygen saturation | 1 minute
  Represented by the microcirculation variables
oxygenated hemoglobin concentration | 1 minute
  Represented by the microcirculation variables
deoxygenated hemoglobin concentration | 1 minute
  Represented by the microcirculation variables
tissue temperature | 1 minute
  Represented by the microcirculation variables
oxygen flow | 1 minute
  Represented by the microcirculation variables

CONTACTS AND LOCATIONS:
Locations (1):
- Rafael Moura Miranda, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Miranda RM, Cabral Filho JE, Diniz KT, Clough GF, Alves JGB, Lima GMS, Figueredo NPDS, Franca AA, Luna JTB. Effect of Kangaroo Position on microcirculation of preterm newborns: a controlled randomized clinical trial. J Pediatr (Rio J). 2022 Mar-Apr;98(2):196-203. doi: 10.1016/j.jped.2021.05.012. Epub 2021 Aug 26. PMID 34454941